CLINICAL TRIAL: NCT03511976
Title: Adaptive Response to Intervention (RTI) for Students With ADHD
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Death of PI
Sponsor: Florida International University (Other)
Collaborators: University at Buffalo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R305A170532
Record Dates: First submitted 2018-04-18; First posted 2018-04-30 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Central Nervous System Stimulants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Business as Usual (BAU) (No Intervention): One-third of participants will be assigned to this condition and will receive academic accommodations and interventions as deemed appropriate by their teachers, school personnel, and parents. This condition is intended to mirror current standard procedures for youth with ADHD. Thus, the specific accommodations and interventions are expected to vary across students. Some students' parents and physicians may choose to start stimulant medication with a goal of improving classroom performance.
- Response to Intervention (RTI): Tier 1 (Experimental): Two-thirds of participants will be assigned to the RTI Tier 1 Arm. Teachers of students in this arm will receive consultation in RTI Tier 1 Classroom Management strategies.
  Interventions: Behavioral: Tier 1 Classroom Management
- RTI: Daily Report Card (DRC) (Experimental): Students assigned to the RTI Tier 1 Arm, who do not respond to the initial RTI Tier 1 Classroom Management strategies, will move to the RTI DRC Arm of the study. Teachers of students in this arm of the study will receive consultation to implement a daily report card.
  Interventions: Behavioral: Tier 1 Classroom Management; Behavioral: Daily Report Card (DRC)
- RTI: Enhanced (Experimental): Half of students in the RTI DRC Arm who do not respond to the DRC intervention will be randomly assigned to the RTI: Enhanced Arm. Students in this arm will receive a more intensive classroom behavioral intervention directed at individual target behaviors through an enhanced DRC.
  Interventions: Behavioral: Tier 1 Classroom Management; Behavioral: Daily Report Card (DRC); Behavioral: Enhanced DRC (DRC-E)
- Medication (Experimental): Half of students in the RTI DRC Arm who do not respond to the DRC intervention will be randomly assigned to the Medication arm and will receive stimulant medication as an additional intervention.
  Interventions: Behavioral: Tier 1 Classroom Management; Behavioral: Daily Report Card (DRC); Drug: Stimulant

INTERVENTIONS:
Behavioral: Tier 1 Classroom Management — The primary teacher for each participating student will receive consultation related to implementing Tier I management strategies at a classroom level for all students including the target child (see Appendix C). Consultation will be provided by trained study personnel and the strategies will be implemented by the general education teacher (i.e., the end user of the intervention)
  Arms: Medication; RTI: Daily Report Card (DRC); RTI: Enhanced; Response to Intervention (RTI): Tier 1
Behavioral: Daily Report Card (DRC) — Students in the RTI DRC condition will receive Tier II strategies, namely an individualized DRC. Behavioral consultants will meet with teachers to identify appropriate behavioral targets and establish a DRC according to established protocol (see our website for an example http://ccf.fiu.edu/for-families/resources-for-parents/printable- information/). Consultants will also meet with parents to develop a plan for reinforcing the DRC at home using a hierarchical menu of rewards/privileges that will be provided contingent on meeting daily goals.
  Arms: Medication; RTI: Daily Report Card (DRC); RTI: Enhanced
Behavioral: Enhanced DRC (DRC-E) — In this condition, students who did not show sufficient response to the Phase 1 DRC will receive additional and more intensive Tier II supports.
  Following student assignment to RTI-E, the teacher will have meet with one of the consultants to complete a functional behavior analysis (FBA) to identify remaining target behaviors and ascertain their function. The consultant and teacher will then use the completed FBA to develop a treatment plan for an enhanced DRC (DRC-E).
  Tier II enhancements will be chosen to directly map on to the functions of the target behaviors as outlined in the FBA.
  Arms: RTI: Enhanced
Drug: Stimulant — Students will receive either a long-acting methylphenidate preparation or a long-acting mixed amphetamine salts preparation based on parent consultation with the study physician. The prescribed medication will be taken daily.
  Other Names: long-acting methylphenidate, long-acting mixed amphetamine salts
  Arms: Medication

SUMMARY:
Purpose: The primary purpose of the proposed project is to investigate the efficacy of Tier 1 and Tier 2 interventions delivered through a Response to Intervention (RTI) framework for children with attention-deficit/hyperactivity disorder (ADHD). Further, for children who do not respond to initial Tier 2 strategies, the proposed study will assess which additional course of intervention is most effective: (1) enhanced Tier 2 strategies or (2) stimulant medication. The majority of youth with ADHD are in general education settings, whether classified as special education students or not. Thus, experimentally evaluating the efficacy of well-developed and evidence-based behavioral interventions within a problem-solving framework such as RTI would significantly inform practice within school-based behavioral intervention teams.

Project Activities: This study will employ a sequential multiple assignment randomized trial design (SMART). Prior to the beginning of the academic year, students will be randomly assigned to one of two conditions: (1) Business as Usual in which children receive whatever sequence of academic supports and interventions their teachers, school, and parents would typically put into place throughout the entire academic year and (2) an RTI approach to begin with Tier 1 classroom-wide management strategies with opportunities to add Tier 2 strategies for youth who do not respond to the initial Tier 1 approach.

DETAILED DESCRIPTION:
Setting: The proposed investigation will be conducted in elementary schools throughout the Western New York and Southern Florida areas.

Sample: Participants will be 300 children, grades 1 - 5, with ADHD who have not been classified as special education students (e.g., Specific learning Disability, Emotional Disturbed, Other Health Impaired), who are not currently prescribed psychoactive medication and are naïve to psychoactive medication. Half of the participants will be recruited in Florida and half will be recruited in New York. This sample is selected to represent school-age children with ADHD who are at elevated risk for referral for special education services.

Intervention: The intervention under study will be a RTI approach for child behavior. The entire intervention includes Tier 1 classwide-behavioral management strategies used by the teacher, a Daily Report Card (DRC) that targets the child's behaviors needed to promote successful social and academic outcomes, and if needed, an enhanced RTI. Participants assigned to the enhanced RTI arm will receive a DRC enhanced with additional behavior management strategies (e.g., differential attention, delayed punishments to reduce escape-maintained behaviors, premack contingencies, etc.) targeting behaviors as indicated by a functional behavior analysis. Participants assigned to the stimulant medication condition will continue to receive the DRC established previously and will also receive stimulant medication during the school day.

Research Design and Methods: One-third of children will be allocated to the BAU condition and two-thirds will be allocated to the RTI approach (Phase 1 Randomization). Children assigned to the RTI approach who do not respond to the Tier 1 strategies will receive a Tier 2 intervention, namely a daily report card (DRC; Phase 2). Children who demonstrate non-response to the DRC will be randomly assigned to one of two additional treatment arms: (1) enhanced RTI (RTI-E) or (2) stimulant medication (Phase 3 Randomization). Children will be allocated evenly across these two conditions.

Control Condition: The RTI framework will be compared with other alternative intervention approaches that represent the standard of care for ADHD treatment in schools (i.e., medication, business as usual classroom intervention) to determine whether this specific model/framework of intervention is efficacious relative to an ecologically valid, counter-factual, comparison group.

Key Measures: Measures of key outcomes will include risk of referral to special education as measured by functional academic outcomes, observations of behavior in the classroom by observers unaware of study hypothesis or treatment condition, and parent and teacher ratings of functioning. Secondary outcome measures will include potential mediators and moderators of treatment response including: discipline referrals, parent contacts due to problems in academic or behavioral functioning, teacher adherence to Tier 1 and Tier 2 strategies, and referrals for an IEP or 504 plan.

Data Analytic Strategy: Specific aims will be addressed using primary data analysis strategies for SMART trials. Specifically, each of the outcome measures will be subjected to the following primary analyses:

Main effect of Phase 1 randomization. Regressions with group membership as a predictor will be used to determine the effect of randomizing participants to either (a) the RTI problem-solving framework approach or (b) business as usual.

Main effect of Phase 3 randomization. Regressions with group membership as a predictor will be used to determine the effect of randomizing non-responders to both Tier 1 classroom management strategies and Tier 2A basic RTI to either (a) enhanced RTI or (b) medication management.

Pairwise comparisons of the three embedded treatment protocols. This SMART design has three embedded treatment protocols, or sets of decision rules that together define an adaptive intervention. Those three protocols are as follows:

1. Business as usual (BAU)
2. Tier 1 strategies, followed by Tier II strategies in the event of non-response (i.e., a DRC), followed by enhanced RTI in the event of non-response.
3. Tier 1 strategies, followed by Tier II strategies in the event of non-response, followed by medication management in the event of non-response

ELIGIBILITY:
Inclusion Criteria:

* Child meets DSM-V diagnostic criteria for Attention-Deficit/Hyperactivity Disorder
* Child will be entering grades 1 - 5

Exclusion Criteria:

* Child or sibling living in the same home has history of sustained successful treatment of ADHD with stimulant medication
* Child currently has a special education placement involving placement in reduced ratio classroom or having a part or full-time aid due to behavior problems
* Child has an IQ less than 70
* Child has psychosis or a pervasive developmental disorder
* Child is in a classroom that already has a study participant
* Child is home-schooled

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2023-10-21 (Actual); Study Completion 2023-10-21 (Actual)

PRIMARY OUTCOMES:
Observations of Classroom Behavior | End of academic year 1 of enrollment
  Independent observations will be conducted using the Student-Behavior Teacher-Response observation system (SBTR; Pelham, Greiner, & Gnagy, 2008; Vujnovic, Fabiano et al., 2014). The SBTR is an observation code that collects information on: (1) the frequency of student rule violations; (2) whether a teacher observed the misbehavior; (3) if observed, whether the teacher enacted a consequence and whether it was an appropriate consequence. The SBTR system also records the number of praise statements and commands issued. The SBTR is a well-defined and validated observation system for use with children with ADHD in classroom settings. The SBTR system documents child functioning across a number of disruptive behavior categories (e.g., be respectful, obey adults, work quietly, stay on task), and it is consistent with an evidence-based assessment procedure for ADHD (Pelham, Fabiano, & Massetti, 2005).

SECONDARY OUTCOMES:
Disruptive Behavior Disorders Rating Scale | End of academic year 1 of enrollment
  Teachers will complete ratings of student classroom behavior
Impairment Rating Scale | End of academic year 1 of enrollment
  Teacher rating of student impairment

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Florida International University Center for Children and Families, Miami, Florida
  - Center for Children and Families, University at Buffalo, Buffalo, New York